CLINICAL TRIAL: NCT01077219
Title: Study on Energy Cost Prediction of Cycle Ergometer
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Ying-Tai Wu, School and Graduate Institute of Physical Therapy, College of Medicine, National Taiwan University
Other Study IDs: 200905044R
Record Dates: First submitted 2010-02-25; First posted 2010-03-01 (Estimated); Last update posted 2010-03-01 (Estimated); Status verified 2010-02

CONDITIONS: Healthy; Obesity
Keywords: healthy female
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study purpose is (1) to develop the new energy expenditure equation; (2) to increase accuracy of energy cost prediction of cycle ergometer; (3) to find out some dependent factors.

DETAILED DESCRIPTION:
Oxygen consumption (ml/min) was measured while subjects were at rest and exercised at four submaximal workloads in steady state on cycle ergometer. Bioelectrical impedance analysis was used to estimate the body fats and skeletal muscle mass.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female
* Never received bicycle training

Exclusion Criteria:

* Exercise testing contraindications

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy female
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Tai Wu, Assoc Prof, Study Chair — School and Graduate Institute of Physical Therapy, College of Medicine, National Taiwan University